CLINICAL TRIAL: NCT02767843
Title: Pilot Study to Assess the Effectiveness and Safety of Continuous Negative External Pressure (cNEP) in Reducing Respiratory Sounds in Individuals With Chronic Snoring
Brief Title: Pilot Study of cNEP for the Treatment of Snoring
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruiting sufficient number of qualified subjects proved impossible.
Sponsor: Sommetrics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOM-011
Record Dates: First submitted 2016-05-09; First posted 2016-05-10 (Estimated); Results first posted 2017-03-24 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-04

CONDITIONS: Snoring
MeSH Terms: conditions — Snoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- treatment (Experimental): continuous negative external pressure (cNEP) at various negative pressures
  Interventions: Device: continuous negative external pressure (cNEP)

INTERVENTIONS:
Device: continuous negative external pressure (cNEP) — soft silicone collar placed on the anterior neck, to which a negative pressure is introduced

SUMMARY:
This pilot study will examine the efficacy and safety of continuous negative external pressure ("cNEP") for the treatment of chronic snoring in people without obstructive sleep apnea.

ELIGIBILITY:
Inclusion Criteria:

* sleep test within the previous six months that shows snoring of at least 30 dB for at least 30% of total sleep time
* AHI < 10/hr

Exclusion Criteria:

* previous neck surgery or radiation
* carotid artery disease
* serious medical or psychiatric illness
* pregnancy
* silicone allergy
* excessive use of alcohol or sedating drugs

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-05; Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerrold Kram, MD, Principal Investigator — California Center for Sleep Disorders, Alameda, CA
Locations (1):
- California Center for Sleep Disorders, Alameda, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Subjects: Only four subjects completed the study.
Period: Overall Study
Arm/Group | Subjects
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: all subjects who underwent cNEP usage
Arm/Group | Treatment
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 42 [33 to 57]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Response
Description: snoring decreased by <50% from baseline
Time Frame: one night
Population: Technical problems with the measurement instruments meant that no analyzable data were collected.
Groups:
- Subjects: Only four subjects were entered into the study. None had outcome measure (2) collected because of technical problems with data collection. Thus no interpretable data were collected.
Arm/Group | Subjects
Number analyzed (Participants) | 0

2. Primary Outcome: Adverse Events
Description: all adverse events
Time Frame: one night
Population: All four participants were analyzed for adverse events. No participants could be analyzed for efficacy outcomes because of technical difficulties with the measurement instruments.
Measure: Count of Participants; unit: Participants
Groups:
- Subjects: Only four subjects were entered into the study.
Arm/Group | Subjects
Number analyzed (Participants) | 4
Participants | 1

3. Secondary Outcome: Complete Response
Description: snoring for < 5% of total sleep tim
Time Frame: one night
Population: Insufficient enrollment to permit analysis.
Groups:
- Subjects: Only four subjects were entered into the study. No efficacy data could be analyzed because of technical problems with the data collection equipment.
Arm/Group | Subjects
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: entire study duration
Groups:
- All Subjects: Only four subjects completed the study.
Arm/Group | All Subjects
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 1/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects (N=4)
minor erythema (Skin and subcutaneous tissue disorders) | 1 (1) — minor erythema, spontaneously resolved

LIMITATIONS AND CAVEATS:
Early termination due to difficulty of recruitment. Technical problems with measurements, so data were uninterpretable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No